CLINICAL TRIAL: NCT02528266
Title: Open Non-randomized Clinical Investigation to Evaluate the Safety and Effectiveness of the Nerve Capping Device to Prevent Neuroma Formation After Traumatic Nerve Section
Brief Title: Surgical Treatment of Symptomatic Neuroma "Stop Neuroma"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polyganics BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 034A01_CIP
Record Dates: First submitted 2015-08-13; First posted 2015-08-19 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Neuroma
MeSH Terms: conditions — Neuroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nerve Capping Device (Experimental): Implant with the experimental device
  Interventions: Device: Nerve Capping Device

INTERVENTIONS:
Device: Nerve Capping Device

SUMMARY:
This study is conducted to clinically assess safety and performance of the Polyganics nerve capping device for the treatment of symptomatic neuroma. There is sufficient clinical experience with regard to the safety of the commercially available nerve guide, NEUROLAC®. This new nerve capping device is identical in material and manufacturing. The exception is in design, where NEUROLAC® has two open ends, the nerve capping device has one closed (sealed) end. This study will be conducted to obtain data on the clinical performance of the capping device's ability to isolate the nerve end, resulting in a reduction of pain of experienced from the symptomatic neuroma and prevention of the reoccurrence of a symptomatic neuroma.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible according to the following criteria:

1. Subjects who are able to provide a written informed consent prior to participating in the clinical investigation.
2. Subjects who are > 18 years year old.
3. Subjects with a diagnosis of symptomatic primary or secondary end-neuroma.
4. Symptomatic neuroma located on the upper limb between the metacarpophalangeal (MCP) joints to shoulder.
5. Symptomatic neuroma confirmed by pain relief following a 10min ±2min nerve block with Xylocaine (Lidocaine) - Pain relief defined as any reduction in VAS questionnaire score.
6. Subjects with history of pain in the area of the end-neuroma for at least 6-months.
7. Subjects with a positive Tinel's sign.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation:

1. Inability to comply with the clinical investigation follow-up or other clinical investigation requirements.
2. Subjects who are pregnant or intend to become pregnant during the duration of the clinical investigation or subjects who are not using appropriate birth control.
3. Subjects who have had historical radiotherapy in the area of the end-neuroma.
4. Symptomatic neuroma located proximally from the shoulder or distally from MCP joints.
5. Subjects not willing to follow post-surgery protocols (e.g. avoiding pressure on the implant zone).
6. Subjects is involved in another pain study.
7. Subjects who have a known allergy to anesthetic agent or bioresorbable copolyester Poly(68/32[15/85 D/L] Lactide-Ԑ-Caprolactone) (PLCL).
8. Subjects with a symptomatic neuroma that underwent surgical treatment for pain management on two or more occasions.
9. Insufficient soft tissue at the end-neuroma site to cover the investigational device.
10. Immunosuppressed patients, or patients with planned immunosuppressive therapy within 12-month following the study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Safety data (Serious adverse events ) | 6 weeks
  Serious adverse events related to the investigation device as determine by independent expert.
Effectiveness (VAS score) | 6 weeks
  Pain caused by symptomatic end-neuroma: VAS score (0-100 / no pain - unbearable pain) at 6-week follow-up compared to score at baseline.
Effectiveness (QuickDASH score) | 6 weeks
  Pain caused by symptomatic end-neuroma: QuickDASH score (30 items scored 1-5) at 6-week follow-up compared to score at baseline.
Effectiveness (Quantity and class of pain medication used) | 6 weeks
  Quantity and class of pain medication used for the end-neuroma pain at 6-week follow-up compared to baseline

SECONDARY OUTCOMES:
Safety (Rate of serious adverse device effects) | 3, 6 and 12 months
  Rate of serious adverse device effects as determined by the physician and independent expert.
  * Reduction of pain caused by symptomatic neuroma after 3 months, 6 months and 12 months following the procedure, as compared to pain before the procedure.
  * Improvement of quality of life at 3 months, 6 months and 12 months follow-up, as compared to the quality of life before the procedure.
  * ≤20% recurrence of symptomatic neuroma within 12 months.
  * Reduction of pain medication used to treat neuroma pain at 3 months, 6 months and 12 months, as compared to the quantity pain medication used for the neuroma pain before the procedure.
Effectiveness (VAS score) | 3, 6, 12 months
  Pain caused by symptomatic end-neuroma: VAS score (0-100 / no pain - unbearable pain) compared to score at baseline.
Effectiveness (QuickDASH score) | 3, 6, 12 months
  Pain caused by symptomatic end-neuroma: QuickDASH score (30 items scored 1-5) compared to score at baseline.
Effectiveness (DN4 score) | 6 weeks, 3, 6, 12 months
  Pain caused by symptomatic end-neuroma: DN4 score (10 y/n items characterising pain) compared to score at baseline.
Effectiveness (Elliot score) | 6 weeks, 3, 6, 12 months
  Pain caused by symptomatic end-neuroma: Elliot score (5 items rated 0 (no pain) to 4 (pain intolerable)) compared to score at baseline.
Effectiveness (Quantity and class of pain medication used) | 3, 6, 12 months
  Quantity and class of pain medication used for the neuroma pain at 3, 6 and 12 months
Rate of recurrence of symptomatic neuroma | 12 months
  defined as daily pain combined with increased used of pain medication compared to baseline and no improvement in QuickDASH score, but pain is relieved with Xylocaine nerve block.

OTHER OUTCOMES:
Usability (User Device Handling Questionnaire) | Day 0
  Ease of placement of the device assessed via User Device Handling Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Betty IJmker, MSc, Study Chair — Polyganics BV
Locations (7):
- Strasbourg University Hospitals, Strasbourg, France
- Netherlands (6):
  - Albert Schweitzer Hospital, Dordrecht
  - UMCG, Groningen
  - Martini Hospital Groningen, Groningen
  - MC Groep, Lelystad
  - MUMC, Maastricht
  - Haga Hospital, The Hague

IPD SHARING:
Plan to Share IPD: Undecided